CLINICAL TRIAL: NCT00618371
Title: Investigating the Source of HIV-1 Viremia in Patients on Antiretroviral Therapy Through Intensification With MK-0518
Brief Title: Pilot Study of Adding Raltegravir (MK-0518) to Antiretroviral Therapy in Patients With Low Level Viremia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Frank Maldarelli, Principal Investigator, National Cancer Institute (NCI)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 27XS050; HHSN261200800001E (Other Grant/Funding Number: SAIC); ZIABC011464 (NIH)
Record Dates: First submitted 2007-09-29; First posted 2008-02-20 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: HIV Infection
Keywords: Intensification; HIV viremia; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir intensification (Experimental): Patients will be administered raltegravir 400 mg orally twice daily in addition to antiretroviral therapy
  Interventions: Drug: Raltegravir (MK-0518)

INTERVENTIONS:
Drug: Raltegravir (MK-0518) — Antiretroviral drug intensification with Raltegravir (MK0518) 400mg orally every 12 hours for 28 days in addition to the prescribed antiretroviral therapy
  Other Names: MK-0518

SUMMARY:
The medicines used to treat HIV can suppress but cannot kill all the virus in the body. A small amount of virus remains at low levels in the part of the blood called the plasma. It is of crucial importance to identify the source of the residual virus in patients receiving antiretroviral therapy. The purpose of this study is to investigate whether the source of low level plasma virus is from latent (old) infection or ongoing (new) infection. MK-0518 is a investigational drug, which means that is not yet FDA approved, that works in a different way to other anti-HIV medicines to help kill the virus. We hypothesize that addition of MK-0518 to a stable anti-HIV regimen will reduce the viral load further in patients with undetectable plasma virus.

DETAILED DESCRIPTION:
This is a non-randomized, non-comparative, single center trial of antiretroviral therapy intensification using the investigational integrase inhibitor MK-0518 and an investigational viral load assay to measure response to additional antiviral therapy. Eighteen patients will receive open-label MK-0518 400 mg P.O. every 12 hours for 28 days in addition to their prescribed antiretroviral therapy. Patients will take their doses of MK-0518 without regard to food. The study will enroll patients on antiretroviral therapy regimens with Cluster of Differentiation 4 (CD4) counts greater than 200 cells/ul, HIV-1 RNA levels <50 copies RNA/ml plasma using a commercial assay(conventional Amplicor) and with detectable plasma virus (viral loads ≥ 1 copies RNA/ml plasma, Single copy assay, "SCA"). Acceptable antiretroviral regimens will include those on Nucleoside reverse transcriptase inhibitors ("NRTIs") + protease inhibitor (PI)I, NRTIs + non-nucleoside reverse transcriptase inhibitors (NNRTIs), + PI, or NRTIs + NNRTI-containing regimens. Patients cannot have prior evidence of resistance to antiretroviral drugs. Patients will be screened for intensification by history, physical exam, and laboratory evaluations (see below). Patients who are eligible and who agree to participate will intensify their antiretroviral therapy for 28 days with MK-0518 400 mg by mouth twice a day. During the 28- day drug addition, patients will have samples drawn for SCA assay at entry and on days 7, 14, 21, and 28 (+/- 1 d), with the last day of intensification as day 28. Patients will have additional phlebotomy after intensification on days 29, 30, 35, 42, 49 and 58 (+/- 1 day). The intensification period is followed by a post- intensification period to determine whether removal of the drug resulted in viral RNA changes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by positive HIV-1 ELISA and positive
* Male or female at least 18 years of age, and able to provide written, informed consent
* Current antiretroviral therapy with Department of Health and Human Services (DHHS)-recommended regimen: NRTIs + PI, NRTIs + NNRTI + PI, or NRTIs + NNRTI
* Screening CD4 > 200 cells/ µl and CD4%> 14%; does not require prophylaxis for opportunistic infections
* Receiving a stable antiretroviral regimen for 4 months prior to screening
* HIV-1 RNA level below the limit of detection by commercial HIV-1 RNA determination assays for at least 12 months prior to screening.
* HIV RNA ≥ 0.6 copy RNA/ml plasma by SCA(single copy assay)
* Hgb ≥ 9.0 mg/dl, absolute neutrophil count > 1000/mm3, platelet count > 100,000/mm3
* Alkaline phosphatase, Aspartate transaminase (AST) and Alanine aminotransferase (ALT) < 2.0 x upper limit of normal
* Willing to take MK-0518 for 28 days in addition to ongoing antiretroviral therapy
* Be considered clinically stable, in the opinion of the investigator, at the time of entry into the study; i.e., clinical status and all chronic medications should be unchanged for at least two weeks prior to entry.

Exclusion Criteria:

* Prior participation in an MK-0518 or other integrase inhibitor trial
* Requires prohibited medications noted in the protocol
* Requires cytotoxic agents including hydroxyurea or vaccinations during the study period
* Received immunosuppressive therapy including steroids within one month prior to treatment in this study
* Used any investigational agents within a month prior to treatment in this study
* Documented resistance to any drug in each of the 4 classes of licensed antiretroviral agents by genotype or phenotype
* Any febrile illness (T>38oC) in the 3 weeks prior to enrollment
* Any vaccination in the 6 weeks prior to enrollment
* Diagnosis of acute hepatitis due to any cause
* Positive Hepatitis B surface antigen
* Severe renal insufficiency defined as a calculated creatinine clearance at time of screening as < 30 ml/min, based on the Cockcroft-Gault equation.
* Condition (including but not limited to alcohol or other substance use) which in the opinion of the investigator would interfere with patient compliance or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah McMahon, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data were analyzed and there is no plan to make individual participant data available

REFERENCES:
- [Background] Natarajan V, Bosche M, Metcalf JA, Ward DJ, Lane HC, Kovacs JA. HIV-1 replication in patients with undetectable plasma virus receiving HAART. Highly active antiretroviral therapy. Lancet. 1999 Jan 9;353(9147):119-20. doi: 10.1016/s0140-6736(05)76156-0. No abstract available. PMID 10023903
- [Background] Dornadula G, Zhang H, VanUitert B, Stern J, Livornese L Jr, Ingerman MJ, Witek J, Kedanis RJ, Natkin J, DeSimone J, Pomerantz RJ. Residual HIV-1 RNA in blood plasma of patients taking suppressive highly active antiretroviral therapy. JAMA. 1999 Nov 3;282(17):1627-32. doi: 10.1001/jama.282.17.1627. PMID 10553788
- [Background] Zhang L, Ramratnam B, Tenner-Racz K, He Y, Vesanen M, Lewin S, Talal A, Racz P, Perelson AS, Korber BT, Markowitz M, Ho DD. Quantifying residual HIV-1 replication in patients receiving combination antiretroviral therapy. N Engl J Med. 1999 May 27;340(21):1605-13. doi: 10.1056/NEJM199905273402101. PMID 10341272
- [Background] Palmer S, Wiegand AP, Maldarelli F, Bazmi H, Mican JM, Polis M, Dewar RL, Planta A, Liu S, Metcalf JA, Mellors JW, Coffin JM. New real-time reverse transcriptase-initiated PCR assay with single-copy sensitivity for human immunodeficiency virus type 1 RNA in plasma. J Clin Microbiol. 2003 Oct;41(10):4531-6. doi: 10.1128/JCM.41.10.4531-4536.2003. PMID 14532178
- [Background] Maldarelli F, Palmer S, King MS, Wiegand A, Polis MA, Mican J, Kovacs JA, Davey RT, Rock-Kress D, Dewar R, Liu S, Metcalf JA, Rehm C, Brun SC, Hanna GJ, Kempf DJ, Coffin JM, Mellors JW. ART suppresses plasma HIV-1 RNA to a stable set point predicted by pretherapy viremia. PLoS Pathog. 2007 Apr;3(4):e46. doi: 10.1371/journal.ppat.0030046. PMID 17411338
- [Background] Hazuda DJ, Wolfe AL, Hastings JC, Robbins HL, Graham PL, LaFemina RL, Emini EA. Viral long terminal repeat substrate binding characteristics of the human immunodeficiency virus type 1 integrase. J Biol Chem. 1994 Feb 11;269(6):3999-4004. PMID 8307956
- [Derived] McMahon D, Jones J, Wiegand A, Gange SJ, Kearney M, Palmer S, McNulty S, Metcalf JA, Acosta E, Rehm C, Coffin JM, Mellors JW, Maldarelli F. Short-course raltegravir intensification does not reduce persistent low-level viremia in patients with HIV-1 suppression during receipt of combination antiretroviral therapy. Clin Infect Dis. 2010 Mar 15;50(6):912-9. doi: 10.1086/650749. PMID 20156060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was approved in 10/2007. HIV-infected individuals 18 years of age receiving stable, suppressive antiretroviral therapy (ART) with persistent plasma HIV-1 RNA level of > 0.6 copies/mL by single-copy assay at screening; enrollment started in in 12/2007 at the University of Pittsburgh Clinical Trials Unit from 12/2007 through 1/2009.
Pre-assignment Details: Participants had Cluster of Differentiation 4(CD4) counts of greater than 200 cells/microliter, HIVRNA< 50 copies/mL plasma for ≥12 months; and not receiving prophylaxis for opportunistic infections (OI)s; no history of exposure to raltegravir, HIV-1 drug resistance,febrile illness within 3 weeks or vaccination within 6 weeks before enrollment.
Groups:
- Group 1: group to be treated with raltegravir
Period: Overall Study
Arm/Group | Group 1
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group receiving raltegravir
Arm/Group | Group 1
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 45.5 (10.6)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HIV-1 RNA Response: ≥ 1 Log Decrease in Viral Load
Description: HIV RNA levels were determined with a non-commercial, sensitive single copy assay for HIV. The primary outcome measure was to determine the number of individuals with ≥10fold decrease in HIV RNA
Time Frame: 4 weeks
Population: Number of participants based on estimates of how many will have decreased viral RNA levels. If 10 participants do not have decreased RNA, the number of patients with potential for decrease is <15% of all suppressed patients.
Measure: Number; unit: participants
Groups:
- Raltegravir Intensification: participants received 4 wk raltegravir intensification
Arm/Group | Raltegravir Intensification
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: Proviral DNA Response, HIV-1 Sequence Variation Levels of Cell Associated HIV DNA and Genetic Variation in HIV During Raltegravir Addition in Individuals Who Have Declines in HIV
Description: We planned to compare HIV DNA levels and HIV genetic variation in individuals with and without ≥10 fold decreases in HIV RNA. As none of the patients had a decline in viral RNA, this analysis could not be readily analyzed
Time Frame: 4 weeks
Population: 0 participants were analyzed because no patients had ≥10 fold decrease in viral RNA. As described in patient outcome description, we would sequence patients only if a ≥10- fold decrease in viremia occurred, Since no one experienced ≥10 fold decrease in viremia, no sequencing could be performed.
Groups:
- Raltegravir Intensification: participants received 4 wk raltegravir intensification. Samples from 0 participants were analyzed No Patients experienced ≥ 1 log decline in viral RNA, so no samples could be analyzed
Arm/Group | Raltegravir Intensification
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: entire trial period of 18 months and thought the end of study period directly after 18 months
Groups:
- Group 1: group treated with raltegravir
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No